CLINICAL TRIAL: NCT04430283
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of Intravenous FDY-5301 for the Prevention and Treatment of ICU Acquired Weakness in Major Trauma Patients.
Brief Title: Evaluation of FDY-5301 in Major Trauma Patients in ICU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated because of difficulty identifying patients that met the inclusion criteria, as well as logistical difficulties in opening clinical ICU study sites.
Sponsor: Faraday Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FDY-5301-203
Record Dates: First submitted 2020-04-20; First posted 2020-06-12 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: ICU Acquired Weakness
Keywords: ICU acquired weakness, PICS, SIRS; Muscle wasting and weakness; muscle function; quality of life
MeSH Terms: conditions — Muscular Atrophy; Asthenia

STUDY DESIGN:
Intervention Model Description: All subjects who fulfill all study edibility criteria will be randomized to receive one of the 3 treatments.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study where all study staff and participants are blinded to whether the patient receives active drug or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FDY-5301 Low Dose (1 mg/kg) (Experimental): FDY-5301 will be administered intravenously once daily for up to 7 days. Dosage will be determined on a body weight basis, according to treatment assignment and using the subject's body weight (estimated or actual) determined at screening.
  Interventions: Drug: FDY-5301
- FDY-5301 High Dose (2 mg/kg) (Experimental): FDY-5301 will be administered intravenously once daily for up to 7 days. Dosage will be determined on a body weight basis, according to treatment assignment and using the subject's body weight (estimated or actual) determined at screening.
  Interventions: Drug: FDY-5301
- Placebo (Placebo Comparator): Placebo will be administered intravenously once daily for up to 7 days. Dosage will be determined on a body weight basis, according to treatment assignment and using the subject's body weight (estimated or actual) determined at screening.
  Other Names:
  Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FDY-5301 — FDY-5301 is Sodium Iodide administered as an isotonic solution for intravenous injection with a concentration of 7.2 mg/ml.
  Arms: FDY-5301 High Dose (2 mg/kg); FDY-5301 Low Dose (1 mg/kg)
Other: Placebo — Placebo is delivered as a single dose, non-reserved liquid parenteral consisting of a formulation matched compendial saline.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics (PK) of FDY-5301 compared to placebo in major trauma ICU patients at risk of intensive care unit acquired weakness (ICUAW)

DETAILED DESCRIPTION:
The purpose of the trial is to evaluate the efficacy, safety, and PK of FDY-5301 compared to placebo in trauma ICU patients at risk of ICUAW.

Muscle wasting occurs rapidly after major trauma and is often associated with multi-organ failure lasting from a few weeks to a long term disability. It is believed that FDY-5301 may help prevent or treat muscle weakness and organ dysfunction in major trauma patients.

Approximately 252 subjects will be randomized (1:1:1) to receive up to 7 daily bolus IV doses of FDY-5301 at 1 mg/kg or 2 mg/kg, or volume-matched placebo. To ensure equal representation in each group, the randomization will be stratified by the presence or absence of any pelvic or lower limb fractures.

All subjects who satisfy the eligibility criteria will be randomly allocated to one of three treatment groups (FDY-5301 low dose, FDY-5301 high dose, or placebo).

All subjects will be followed for 6 months.

This study will be conducted globally.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Major trauma defined as:

   1. thoracic and/or abdominal and/or pelvic injury
   2. necessitating admission to ICU with ventilation anticipated for at least 24 hrs
   3. hemorrhagic shock defined as systolic blood pressure (SBP) <90 mmHG requiring blood transfusion or base deficit of at least 6mEq/L pre-hospital arrival or within one hour after hospital arrival
3. IRB/IEC-approved consent obtained within 48 hours of first hospital arrival time (i.e., in case of transfers, use time of arrival to first hospital immediately post injury)

Exclusion Criteria:

1. Likely to die within 48 hrs from time of screening
2. Any neurological condition that is perceived at the time of hospital admission as an immediate threat to life or incompatible with good functional recovery and where early limitation or withdrawal of therapy is being considered. For example:

   a. Computed tomography imaging showing evidence of traumatic brain injury (TBI), combined with best representative Glasgow Coma Score (GCS) Motor Score of ≤4 at approximately 24 hrs post injury
3. Evidence of nonreversible spinal cord injury
4. Bilateral femoral fractures
5. Women who are pregnant or breastfeeding. Women of reproductive potential must have a negative serum pregnancy test prior to randomization.
6. Known thyroid disease or thyroid disorder, including subjects on thyroid hormone replacement therapy at the time of randomization
7. Known allergy to iodine
8. Chronic renal disease requiring dialysis
9. Body mass index (BMI) >40 kg/m2 or <16 kg/m2
10. Body weight (BW) >140 kg (or >309 lb)
11. History or presence of debilitating neurologic or other neuromuscular disease (e.g., spina bifida, amyotrophic lateral sclerosis, multiple sclerosis) at time of randomization
12. Current metastatic cancer
13. Solid organ transplant recipient
14. Evidence of pre-existing sarcopenia defined as having a pre-trauma Clinical Frailty Score (CFS) of ≥5 or based on clinical judgement (e.g. frail by appearance, cachexia, etc.)
15. Use of systemic corticosteroids, immunomodulators, or oncologic chemotherapy within 6 months of randomization (inhaled and topical steroids are allowed)
16. Use of investigational drugs or devices within 30 days of randomization
17. Any clinically significant abnormality identified prior to randomization that in the judgment of the Investigator or Sponsor would preclude safe completion of the study, or confound the anticipated benefit of FDY-5301

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Massachusetts General Hospital, Harvard Medical School, Boston, Massachusetts
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Harborview, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- FDY-5301 Low Dose: 1 mg/kg FDY-5301 will be administered intravenously once daily for up to 7 days.
- FDY-5301 High Dose: 2 mg/kg FDY-5301 will be administered intravenously once daily for up to 7 days.
- Placebo: Placebo will be administered intravenously once daily for up to 7 days.
Period: Overall Study
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo
Started | 2 | 2 | 4
Completed | 0 | 0 | 0
Not Completed | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4 | 8
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34 [29 to 39] | 32.5 [32 to 33] | 25.25 [22 to 30] | 29.25 [22 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 2 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 2 | 3 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Chelsea Critical Care Physical Assessment Tool
Description: Chelsea Critical Care Physical Assessment Tool (CPAx) total score at Day 10, or hospital discharge, whichever occurs first. The Chelsea Critical Care Physical Assessment Tool components will be graded on a 6-point scale from dependent to independent (0 to 5). The individual values will be collated giving a total score out of 50. A higher score indicates a better outcome.
Time Frame: Day 10 or hospital discharge, whichever occurs first.
Population: Overall number of participants analyzed for CPAx data includes only those who have Day 10 CPAx scores. The small number of subjects enrolled in each of the groups preclude interpretation of the CPAx data.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 1 | 2 | 3
Score on a scale | 9 [lower limit 9] | 31.5 [28 to 35] | 11 [10 to 12]

2. Primary Outcome: Organ Dysfunction Total Time to Recovery
Description: Organ dysfunction total time to recovery (TTR) until Day 28
Time Frame: Day 28 or hospital discharge, whichever occurs first.
Population: The small number of subjects enrolled in each of the groups preclude interpretation of the organ dysfunction total TTR data.
Measure: Mean (Full Range); unit: Days
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 2 | 2 | 4
Days | 8.5 [5 to 12] | 4 [2 to 6] | 6 [4 to 8]

3. Secondary Outcome: Medical Research Council Sum Score
Description: Medical Research Council Sum Score (MRC-SS) at Day 28, or hospital discharge, whichever occurs first. The Medical Research Council Sum Score measures global peripheral muscle strength which ranges from 0 (complete paralysis) to 60 (normal strength). A higher score indicates a better outcome.
Time Frame: Day 28, or hospital discharge, whichever occurs first
Population: The small number of subjects enrolled in each of the groups preclude interpretation of the MRC-SS data.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 1 | 0 | 2
Score on a scale | 20 [lower limit 20] |  | 31.5 [15 to 48]

4. Secondary Outcome: Sequential Organ Failure Assessment Score
Description: The Sequential Organ Failure Assessment (SOFA) is a scoring system that assesses the performance of several organ systems in the body and assigns a score based on the data obtained in each category, this is scored during the ICU stay. The full-length Sequential Organ Failure Assessment score ranges from 0 to 24. A higher score indicates a worse outcome.
Time Frame: ICU hospital stay until Day 28 or ICU discharge if earlier
Population: The small number of subjects enrolled in each of the groups preclude interpretation of the SOFA data.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 2 | 2 | 4
Score on a scale | 7.5 [6 to 9] | 6.5 [6 to 7] | 7.5 [4 to 11]

5. Secondary Outcome: Overall Survival at Day 28
Description: Confirmation of survival status will be obtained by speaking directly with subject, via medical records, or public health records.
Time Frame: Day 28
Population: The small number of subjects enrolled in each of the groups preclude interpretation of the Overall Survival at Day 28 data.
Measure: Count of Participants; unit: Participants
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 2 | 2 | 4
Participants | 2 | 2 | 4

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the time of consent until Day 28 were collected.
Description: All safety measures are summarized descriptively. AEs are summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term.
Arm/Group | FDY-5301 Low Dose | FDY-5301 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDY-5301 Low Dose (N=2) | FDY-5301 High Dose (N=2) | Placebo (N=4)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDY-5301 Low Dose (N=2) | FDY-5301 High Dose (N=2) | Placebo (N=4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyporeflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Faraday agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Faraday supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial through a multi-center publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT04430283/Prot_SAP_001.pdf